CLINICAL TRIAL: NCT00004794
Title: Phase II Randomized Study of Cidofovir for Peripheral Cytomegalovirus Retinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11927; NU-506
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: Cytomegalovirus Retinitis; Acquired Immunodeficiency Syndrome
Keywords: cytomegalovirus retinitis; ophthalmologic disorders; rare disease
MeSH Terms: conditions — Cytomegalovirus Retinitis; Acquired Immunodeficiency Syndrome; Rare Diseases | interventions — Cidofovir

INTERVENTIONS:
Drug: cidofovir

SUMMARY:
OBJECTIVES: I. Evaluate the safety and efficacy of intravenous cidofovir in patients with small peripheral cytomegalovirus retinitis.

II. Obtain safety and efficacy data related to different dosages of cidofovir.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Cidofovir is administered intravenously. Treatment ideally begins within 24 hours of randomization.

In the first group, therapy is deferred until disease progression. Patients are then treated according to best medical judgement, which includes the option of cidofovir therapy.

The second group receives induction with cidofovir every 7 days for 2 weeks, then begins maintenance with a low dose given every 14 days until dose-limiting toxicity or disease progression occurs.

The third group receives the same cidofovir induction followed by a high maintenance dose given every 14 days until dose-limiting toxicity or disease progression occurs.

Probenecid and intravenous hydration are administered concurrently with cidofovir.

Patients are followed for progression and survival every 2 weeks for 23 weeks, then every 12 weeks. At disease progression, patients may be re-treated with another course of induction and maintenance.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Acquired immunodeficiency syndrome (AIDS) Meets Centers for Disease Control and Prevention definition
* Peripheral cytomegalovirus (CMV) retinitis Diagnosed by ophthalmologist certified by the Study of Ocular Complications of AIDS group At least 1 lesion measuring at least 25% of disc on photograph No lesion within zone 1 No lesion involving 25% or more of retina regardless of location
* Visual acuity in affected eye 3 or more lines on the Early Treatment Diabetic Retinopathy Study chart at 1 meter Snellen equivalent 8/200
* No retinal detachment in affected eye
* No media opacity that precludes visualization of fundus in both eyes
* No extraocular CMV disease

--Prior/Concurrent Therapy--

* No prior or concurrent anti-CMV therapy, i.e.: Ganciclovir Foscarnet CMV hyperimmune immunoglobulin Other investigational agents with anti-CMV activity
* Prior CMV prophylaxis allowed
* At least 7 days since nephrotoxic drugs, including: Amphotericin B Vidarabine Aminoglycoside antibiotics Intravenous pentamidine

--Patient Characteristics--

* Age: 13 to 60
* Performance status: Karnofsky 60%-100%
* Hematopoietic: ANC at least 750 Platelets at least 50,000 Hemoglobin greater than 7.5 g/dL
* Hepatic: Bilirubin no greater than 3.0 mg/dL Transaminases no greater than 5 times normal
* Renal: Creatinine no greater than 1.5 mg/dL Proteinuria less than 1+ No clinically significant renal disease No dialysis
* Cardiovascular: No clinically significant cardiac disease, including: Ischemia Congestive heart failure Arrhythmia
* Other:

No probenecid allergy No medical problems sufficient to hinder compliance with therapy or follow- up, including drug or alcohol abuse No pregnant or nursing women Negative serum pregnancy test required of fertile women Adequate birth control required of fertile patients during and for 3 months after study

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 1995-03

CONTACTS AND LOCATIONS:
Overall Officials: David V. Weinberg, Study Chair — Northwestern University